CLINICAL TRIAL: NCT06136169
Title: Reminder-cue Scanning Training for People With Homonymous Visual Field Loss
Brief Title: Reminder-cue Scanning Training for Homonymous Visual Field Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Alexandra Bowers, Associate Scientist, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HST_Pilot; R01EY025677 (NIH)
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Homonymous Hemianopia; Homonymous Quadrantanopia
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- StudyArm (Experimental): Participants will receive reminder-cue scanning training in a driving simulator.
  Interventions: Behavioral: Reminder-cue scanning training

INTERVENTIONS:
Behavioral: Reminder-cue scanning training — Auditory reminders to scan when scanning to the side of the field loss is inadequate

SUMMARY:
This study will evaluate a new approach to training people with visual field loss to scan when driving

DETAILED DESCRIPTION:
Homonymous visual field loss is the loss of vision on the same side in both eyes. The most common types are hemianopia (the loss of one half of the field of vision) and quadrantanopia (the loss of one quarter of the field of vision). Hemianopia and quadrantanopia may cause difficulties in seeing objects on the side of the field loss. People with these types of field loss can compensate by scanning (looking) toward the side of the field loss. However, sometimes they might not scan sufficiently well resulting in delayed responses to hazards when driving. The purpose of this research study is to evaluate a new approach, "reminder-cue scanning training", to training people with homonymous visual field loss to scan when driving.

Participants will receive reminder-cue scanning training in the driving simulator.Typically there will be three training sessions within about a 2-week period. In addition, participants will complete an evaluation in the driving simulator before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Homonymous hemianopia or homonymous quadrantanopia for at least 3 months
* Binocular visual acuity of at least 20/40
* Prior or current driving experience
* Able to attend multiple study visits
* Able to communicate in English sufficiently to understand the study procedures

Exclusion Criteria:

* Physical or general health problems that could impair the ability to operate the controls of the driving simulator or participate in the training

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of early large head scans to the side of the field loss | Pre-training, post-training (1 week)
  Proportion of intersections at which an early large head scan was made to the side of the field loss
Detection rate for hazards on the side of the field loss | Pre-training, Post-training (1 week)
  Proportion of hazards detected out of the total number of hazards on the side of the field loss

SECONDARY OUTCOMES:
Rate of early large head scans to the side of the field loss | Pre-training, post-training (up to 12 months)
  Proportion of intersections at which an early large head scan was made to the side of the field loss
Frequency of head scans to the side of the field loss | Pre-training, Post-training (up to 12 months)
  Number of head scans per intersection to the side of the field loss
Magnitude of head scans to the side of the field loss | Pre-training, Post-training (up to 12 months)
  Mean magnitude (in degrees) of head scans to the side of the field loss
Detection rate for hazards on the side of the field loss | Pre-training, post-training (up to 12 months)
  Proportion of hazards detected out of the total number of hazards on the side of the field loss
Response times to hazards on the side of the field loss | Pre-training, Post-training (up to 12 months)
  Mean time (in seconds) between the hazard appearing and the horn-press response

CONTACTS AND LOCATIONS:
Overall Officials: Alex Bowers, PhD, Principal Investigator — Schepens Eye Research Institute of Mass Eye and Ear
Locations (1):
- Schepens Eye Research Institute of Mass Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No